CLINICAL TRIAL: NCT02993640
Title: Effects of Vasopressin and Nitroglycerine in Combination on Splanchnic Blood Flow, and on Hepatic and Portal Venous Pressures in Liver Resection
Brief Title: Optimization of Hepatic Hemodynamics During Liver Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Ellinor Wisén, MD, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EPN879-13
Record Dates: First submitted 2016-12-12; First posted 2016-12-15 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Portal Blood Pressure; Liver Surgery; Hepatic Hemodynamics
Keywords: vasopressin; nitroglycerine; portal pressure; portal flow
MeSH Terms: conditions — Diabetes Insipidus | interventions — Vasopressins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vasopressin + nitro (Experimental): vasopressin + nitroglycerin in simultaneous infusion
  Interventions: Drug: vasopressin + nitro

INTERVENTIONS:
Drug: vasopressin + nitro — vasopressin infusion 4,8 U/h for 20 minutes, thereafter nitroglycerine infusion to a MAP of 60 for 5 minutes.

SUMMARY:
The purpose of this study is to determine if vasopressin and nitroglycerin in combination will affect hepatic hemodynamics, in the setting of liver surgery.

DETAILED DESCRIPTION:
The patients in this study (undergoing elective liver resection) will be anesthetized according to routine practice in our hospital. A radial arterial catheter and a central venous catheter will be inserted, as well as a femoral arterial catheter for Picco monitoring. After the dissection phase, catheters will be inserted in the portal and hepatic veins by the surgeon. Base line data (HR, CVP, MAP, CO from thermodilution, portal and hepatic venous pressure, blood gases from radial artery, vena cava superior, hepatic vein and portal vein) will be obtained twice, with 10 minutes of steady state in between. An infusion of vasopressin 4,8 U/h will then be started and continued for 20 minutes. Data will be collected again, and an infusion of nitroglycerine (to a target of MAP 60 mmHg) will be added. After 5 minutes of steady MAP 55-65, the last set of data is collected. 12 Patients will be recruited, and the total data collection is estimated to be completed and assessed after six to nine months.

ELIGIBILITY:
Inclusion Criteria:

* Patients within ASA-class I-II scheduled for open liver resection

Exclusion Criteria:

* ASA-class III and IV, more than 2 medications for hypertension, BMI > 35, technical difficulties with insertion av catheters, extensive surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Portal and hepatic venous flow after vasopressin and nitroglycerine infusion | six - nine months
Pressure in the hepatic and portal veins after vasopressin and nitrovasopressin infusion | six - nine months

SECONDARY OUTCOMES:
lactate in the splanchnic circulation | six-nine months

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Erik Ricksten, Professor, Study Director — Sahlgrenska University Hospital

IPD SHARING:
Plan to Share IPD: No
No plans of sharing IPD

REFERENCES:
- [Derived] Wisen E, Svennerholm K, Bown LS, Houltz E, Rizell M, Lundin S, Ricksten SE. Vasopressin and nitroglycerin decrease portal and hepatic venous pressure and hepato-splanchnic blood flow. Acta Anaesthesiol Scand. 2018 Aug;62(7):953-961. doi: 10.1111/aas.13117. Epub 2018 Mar 26. PMID 29578250